CLINICAL TRIAL: NCT01180361
Title: Atherosclerosis in RA and Lupus: Restoring Cholesterol Balance
Brief Title: Atherosclerosis in Rheumatoid Arthritis and Lupus: Restoring Cholesterol Balance
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 19-00931
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; systemic lupus erythematosus; atherosclerosis; adenosine
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Active SLE patients: Age 18-65; female and male. No methotrexate or statin therapy in prior 3 months. Not on biological therapies. Fulfill 1982 ACR revised criteria for SLE. SLE activity status designated using the SLEDAI disease activity index. Patients excluded if previous documentation of a connective tissue disorder other than SLE.
- Psoriatic arthritis: Age 18-65; female and male. No methotrexate or statin therapy in prior 3 months. Not on biological therapies. Diagnosed according to criteria described by McGonagle et al (McGonagle, D., Conaghan, P.G., and Emery, P. Psoriatic arthritis: a unified concept twenty years on. Arthritis Rheum 1999; 42: 1080-1086.)
- Normal controls: Age 18-65; female and male. No methotrexate or statin therapy in prior 3 months. Not on biological therapies. Healthy volunteers. Not on corticosteroids.
- Active RA patients: Age 18-65, male and female, no methotrexate or statin therapy in prior 3 months. Not on biological therapies. satisfy at least 4 of the 7 revised criteria (1987) for the classification of RA

SUMMARY:
Hypothesis: SLE and RA increase risk of myocardial infarction (MI, heart attack). Immune reactants in the circulation of SLE patients downregulate cholesterol efflux proteins 27-hydroxylase and ABCA1 and upregulate scavenger receptor CD36, thus encouraging cholesterol accumulation. Adenosine A2A receptor agonist or statin treatment of cells exposed to SLE plasma (or immune complexes or cytokine-enriched plasma fractions from SLE patients) may ameliorate inflammatory properties of their plasma, lessening its atherogenic potency.

Rationale: SLE and RA plasma contain components not present in significant levels in normal plasma that could, individually or acting together, affect 27-hydroxylase, ABCA1 and CD36 expression. Candidate components include autoantibodies, immune complexes, and various cytokines. Statins reduce major cardiovascular events and death. Modulation of adenosine signaling participates in regulation of 27-hydroxylase and ABCA1. As a potential preventative and therapeutic approach to atherosclerotic cardiovascular disease, the investigators evaluate the effect of A2A receptor agonists and statins on atherogenic parameters in SLE and RA plasma.

Experimental Plan: Quantitate 27-hydroxylase and several other proteins involved in cellular cholesterol uptake and excretion in THP-1 monocytes/macrophages and HAEC after exposure to plasma and plasma components from SLE patients (and controls) ± lipid loading with acetylated LDL with/without addition of A2AR agonist, statin, or both. Determine relative impact of immune complexes and cytokines on expression of proteins involved in cholesterol flux. Determine levels of proteins involved in cellular cholesterol influx/efflux in peripheral blood mononuclear cells isolated from RA, SLE and psoriatic arthritis patients and normal controls at baseline, then following incubation in culture media alone or with statin, adenosine A2A agonist or both statin + A2AR agonist.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease (ASCVD) is a major cause of morbidity and mortality, especially in patients with autoimmune disorders such as systemic lupus erythematosus (lupus) and rheumatoid arthritis (RA). We have found that immune and inflammatory mediators promote atherosclerosis by disabling mechanisms that prevent cells of the artery wall from being overloaded with cholesterol, leading to formation of lipid laden foam cells. This proposal seeks to identify which specific components in the blood of patients with lupus and RA make them vulnerable to ASCVD and to explore potential novel therapeutic approaches utilizing our finding that the naturally occurring anti-inflammatory molecule adenosine can restore normal cholesterol outflow to cells that line the artery wall.

1. A 40 cc blood sample will be taken from each subject by venipuncture. The plasma will be added to cell culture media (25 and 50% vol/vol) and used for incubation with THP-1 monocytic leukemia cells and/or human monocyte-derived macrophages and/or human aortic endothelial cells so that the effect of exposure to various disease and control plasma on cholesterol homeostatic protein expression by the cultured cells can be assessed. PBMC will be isolated from a portion of the sample by Ficoll hypaque gradient centrifugation.

   Subject Inclusion & Exclusion Criteria
   1. Normal Controls Normal healthy volunteers, age 18-65, not on corticosteroids or any other immune-modifying medications. Because SLE is a disease with >90% female prevalence and RA has a similar gender bias towards the female sex, our data in men will be exploratory only and we will not be able to examine sex differences in effects on our outcome measures (1, 2).
   2. Rheumatoid Arthritis Patients Patients age 18-65 who satisfy at least 4 of the 7 revised criteria (1987) for the classification of rheumatoid arthritis (3).
   3. Active SLE patients Patients, age 18-65, must fulfill the 1982 revised criteria of the American College of Rheumatology (formerly the American Rheumatism Association) for classification of SLE (4). SLE activity status will be designated using the SLEDAI disease activity index (5). Patients with previous documentation of a diagnosis of a connective tissue disorder other than SLE will be excluded. Patients will have had no statin treatment in the prior three months.
   4. Psoriatic Arthritis Patients Diagnosed according to criteria described by McGonacle et al (6). Defined as an inflammatory arthritis associated with psoriasis

      40 patients will be recruited for each group. Anti-C1q antibodies will be measured in all subjects by a solid-phase enzyme-linked immunosorbent assay.
2. Protection of Human Subjects- Informed consent will be obtained from all subjects and patient confidentiality will be maintained at all times. The protocol and consent form will be approved by the Winthrop University Hospital IRB. We are not using a case study approach so all data will be pooled and anonymity will be preserved. To further ensure anonymity, all records and blood specimens will be numerically coded, and the translation table will be accessible only to the PI. Patients will be asked by their physicians during routine visits to participate in the study.
3. Sources of research material- Blood sample (40 cc) drawn during routine outpatient visits to the faculty practices offices of Winthrop University Hospital Academic Rheumatologists. Patient charts will be utilized to obtain information on disease activity status, medication regimen, age, sex and cardiovascular disease history. All such information is collected in the patient chart as part of standard medical recordkeeping.
4. Potential Risk to Subjects The studies proposed only require the donation of blood samples (40 cc each) by the subjects and impose only the minimal risk to the subjects of blood drawing. These risks include hematoma formation and, very rarely, infection at the puncture site. No interventions or special measures are involved. Furthermore, as patients with the diagnoses of SLE and RA require frequent monitoring of blood parameters, whether in relation to their disease activity or for monitoring the side effects of the treatments they receive, the acquisition of the blood samples for the study impose no additional discomfort to them than what they would experience in their routine medical care. The course of treatment for the subjects will not be changed in any way by participation in this project. All blood specimens will be handled carefully and with full blood precautions.
5. The Risks of this Study are no more than those involved in any routine blood drawing. Donating blood may occasionally cause pain, bruising, fainting or a small infection at the puncture site.
6. Potential Benefits of the Proposed Research to the Subjects and Others At this time, there is no direct benefit for enrolled subjects. However, we hope to gather information that may help people in the future by reducing morbidity and mortality from cardiovascular disease.
7. The Importance of the Knowledge to Be Gained Although the patients will see no direct personal benefit, the knowledge to be gained has immense potential to benefit SLE and RA patients because it may eventually lead us to an understanding of the role of immunological mechanisms in the pathogenesis of premature cardiovascular disease. This understanding will pave the way for the development of life-prolonging preventive and therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18-65

Exclusion Criteria:

* No methotrexate or statin therapy in prior 3 months.
* Not on biological therapies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lupus patients, rheumatoid arthritis patients, psoriatic arthritis patients, healthy volunteers in Nassau County NY
Sampling Method: Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Comparison of 27-hydroxylase level in THP-1 monocytes incubated in human plasma (RA patient, SLE, normal control, psoriatic arthritis). | 3 years
  The activated proinflammatory state of monocytes in RA and SLE subjects constitutes a novel parameter of risk associated with this disorder, related to altered expression of cholesterol transport genes. 27-hydroxylase level may be diminished by the plasma of patents with autoimmune rheumatic disorders.

SECONDARY OUTCOMES:
Plasma 27-hydroxycholesterol levels. | 3 years
  Plasma 27-hydroxycholesterol may be lower in RA and SLE patients than in healthy controls due to less 27-hydroxylase expression and activity in RA and lupus.

CONTACTS AND LOCATIONS:
Overall Officials: Allison B Reiss, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Hospital - Long Island, Mineola, New York, United States

REFERENCES:
- [Background] Reiss AB. Effects of inflammation on cholesterol metabolism: impact on systemic lupus erythematosus. Curr Rheumatol Rep. 2009 Aug;11(4):255-60. doi: 10.1007/s11926-009-0036-y. PMID 19691928
- [Background] Reiss AB, Anwar F, Chan ES, Anwar K. Disruption of cholesterol efflux by coxib medications and inflammatory processes: link to increased cardiovascular risk. J Investig Med. 2009 Aug;57(6):695-702. doi: 10.2310/JIM.0b013e31819ec3c7. PMID 19289972
- [Result] Reiss AB, Wan DW, Anwar K, Merrill JT, Wirkowski PA, Shah N, Cronstein BN, Chan ES, Carsons SE. Enhanced CD36 scavenger receptor expression in THP-1 human monocytes in the presence of lupus plasma: linking autoimmunity and atherosclerosis. Exp Biol Med (Maywood). 2009 Mar;234(3):354-60. doi: 10.3181/0806-BC-194. Epub 2009 Jan 14. PMID 19144874